CLINICAL TRIAL: NCT02496091
Title: A Retrospective Multicenter Study Evaluating ATLANTIS™ Abutments on Implants From Four Manufacturers
Brief Title: Multicenter Retrospective Study Evaluating ATLANTIS™ Abutment Teeth Connected to Implants
Status: Completed | Type: Observational
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Other Study IDs: C-AA-14-003
Record Dates: First submitted 2015-05-20; First posted 2015-07-14 (Estimated); Results first posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Dental Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- ATLANTIS Abutment: The investigational product (ATLANTIS abutment) is already included in a restoration in the subject at enrollment, thus this study does not involve the installation of any investigational products.
  Interventions: Device: ATLANTIS Abutment

INTERVENTIONS:
Device: ATLANTIS Abutment

SUMMARY:
The study is designed as a retrospective and multi-center study. The study population is US individuals previously restored with titanium and gold-shaded titanium ATLANTIS abutments. The study includes retrospective data collection from the medical records and data collection from one prospective study visit with a clinical examination.The primary objective is to evaluate success. Success is defined as that the study implant and abutment are in situ and no Adverse Device Effects related to the study implant, abutment or adjacent peri-implant tissues are reported during the study.

ELIGIBILITY:
Inclusion Criteria:

* Having received one or more ATLANTIS abutments included in one or more permanent prosthetic restoration(s):

  * during 2010, 2011, 2012 or 2013
  * made of titanium or gold-shaded titanium
  * connected to implants from: BIOMET 3i; Straumann; Nobel Biocare or DENTSPLY Implants (only ASTRA TECH Implant System).
* Being at least 18 years at day of enrollment
* Having signed and dated the informed consent form

Exclusion Criteria:

* Unable to come for study visit
* Not willing to participate in the study or not able to understand the content of the study.
* Involvement in the planning and conduct of the study (applies to both DENTSPLY Implants staff and staff at the study site).
* Simultaneous participation in another clinical study that may interfere with the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is individuals who received ATLANTIS abutments, between 2010 and 2013, connected to implants from BIOMET 3i, Straumann, Nobel Biocare or DENTSPLY Implants (only ASTRA TECH Implant System) replacing one or more teeth, in any position in the mouth, as part of a permanent prosthetic restoration. The partially dentate individuals have received either single-unit crowns or fixed partial or full dentures. The abutments need to be titanium or gold-shaded titanium.
Sampling Method: Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ingeborg J. Dr De Kok, DDS, Principal Investigator — University of North Carolina, School of Dentistry, Chapel Hill, NC 27599, US
Locations (6):
- United States (6):
  - University of Alabama at Birmingham, Division of Prosthodontics, Birmingham, Alabama
  - University of California, Los Angeles, School of Dentistry, Los Angeles, California
  - Nova Southeastern University, College of Dental Medicine, Fort Lauderdale, Florida
  - University of Iowa, College of Dentistry, Iowa City, Iowa
  - Columbia University, College of Dental Medicine, New York, New York
  - University of North Carolina, School of Dentistry, Chapel Hill, North Carolina

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Abutments
Groups:
- ATLANTIS Abutment: ATLANTIS Abutment, component used in permanent dental prosthetic restorations. Used for connecting the dental implant with the dental restoration.
Period: Overall Study
Arm/Group | ATLANTIS Abutment
Started | 144; 263 Abutments
Completed | 142; 259 Abutments
Not Completed | 2; 4 Abutments
Not completed — Eligibility criteria not fulfilled | 2

BASELINE CHARACTERISTICS:
Units Other Than Participants: Abutments
Arm/Group | ATLANTIS Abutment
Number analyzed (Participants) | 142
Number analyzed (Abutments) | 259
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 61
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: Participants]
  United States | 142

OUTCOME MEASURES:

1. Primary Outcome: Overall Success Rate
Description: Success defined as study position implant and abutment in situ and no Adverse Event(s) related to implant, abutment or adjacent peri-implant tissues reported during study.
Time Frame: Minium of 2 years and a maximum of 8 years of use.
Population: 144 subjects (263 implant positions) were signed informed consent and were enrolled in the study. 2 subject (4 implant positions) were excluded due to eligibility criteria not fulfilled.
  As a result, a total of 142 subjects (259 implant positions) are included in the analysis.
Measure: Count of Units; unit: Abutments
Units Other Than Participants: Abutments
Arm/Group | ATLANTIS Abutment
Number analyzed (Participants) | 142
Number analyzed (Abutments) | 259
Abutments | 240
Statistical Analysis 1: Comparison: ATLANTIS Abutment; Only descriptive statistics The implant success rate is analyzed on an implant level (i.e. percent of successful implants) as well as subject level (i.e. percentage of subjects with no unsuccessful implants). This proportion is presented together with a 95% confidence interval (using the exact Binomial approach) and an average follow-up time; Test type: Other; 95% confidence interval (using the exact = 92.7, 95% CI 2-sided [88.8 to 95.5]

2. Secondary Outcome: Study Position Implant and Abutment Survival
Description: Survival defined as study position implant and abutment in situ during study. The presence of the study position implant and abutment in the mouth was recorded. The implant and abutment had to be the ones included in the permanent prosthetic restoration when it was delivered / installed.
  Each study position was categorized as survived (No/Yes). It was categorized as survived=Yes when both had been in situ during study. It was categorized as survived=No when either the implant or abutment had been lost during study.
Time Frame: Minium of 2 years and a maximum of 8 years of use.
Population: 144 subjects (263 implant positions) were enrolled in the study. 2 subject (4 implant positions) were excluded due to eligibility criteria not fulfilled giving a per protocol population of 142 subjects (259 positions).
Measure: Count of Units; unit: Abutments
Units Other Than Participants: Abutments
Groups:
- ATLANTIS Abutment: ATLANTIS Abutment, component used in permanent dental prosthetic restorations.
Arm/Group | ATLANTIS Abutment
Number analyzed (Participants) | 142
Number analyzed (Abutments) | 259
Abutments | 256

3. Secondary Outcome: Presence of Plaque
Description: Presence of plaque was evaluated at four surfaces around each study position (mesial, facial, distal and lingual). Plaque was recorded as presence or absence of plaque by visual inspection.
Time Frame: Minium of 2 years and a maximum of 8 years of use.
Population: 144 subjects (263 implant positions) were enrolled in the study. 2 subject (4 implant positions) were excluded due to eligibility criteria not fulfilled giving a per protocol population of 142 subjects (259 positions) .
  Plaque assessment was not completed for 4 positions. As a result, a total of 255 positions are included in the Plaque analysis.
Measure: Count of Units; unit: Positions
Units Other Than Participants: Positions
Arm/Group | ATLANTIS Abutment
Number analyzed (Participants) | 140
Number analyzed (Positions) | 255
Positions | 96

4. Secondary Outcome: Evaluation of the Periimplant Mucosa Condition - By Assessment of PPD
Description: PPD was evaluated at four surfaces around each study position (mesial, facial, distal and lingual), using a periodontal probe. PPD was measured as the distance from the mucosal margin to the bottom of the probeable pocket in whole millimetre. PPD mean values per study positon were calculated.
Time Frame: Minium of 2 years and a maximum of 8 years of use.
Population: 144 subjects (263 implant positions) were enrolled in the study. 2 subject (4 implant positions) were excluded due to eligibility criteria not fulfilled giving a per protocol population of 142 subjects (259 positions) .
  PPD assessment was not completed for 4 positions. As a result, a total of 255 positions are included in the PPD analysis.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Position
Arm/Group | ATLANTIS Abutment
Number analyzed (Participants) | 140
Number analyzed (Position) | 255
Millimeter | 3.11 (1.00)

5. Secondary Outcome: Evaluation of the Periimplant Mucosa Condition - By Assessment of BoP
Description: Condition of the periimplant mucosa by assessment of Bleeding on Probing (BoP). BoP was evaluated at four surfaces around each study position (mesial, facial, distal and lingual), using a periodontal probe.
  BoP was recorded as presence or absence of bleeding when probing to the bottom of the pocket. Presented as % of positions that show presence of bleeding on probing at time of the follow-up visit.
Time Frame: Minium of 2 years and a maximum of 8 years of use.
Population: as for outcome 4
Measure: Count of Units; unit: Positions
Units Other Than Participants: Positions
Arm/Group | ATLANTIS Abutment
Number analyzed (Participants) | 140
Number analyzed (Positions) | 255
Positions | 124

6. Secondary Outcome: Marginal Bone Level Change
Description: Marginal bone level (MBL) determined from radiographs and expressed as the distance from a reference point on the implant to the most coronal bone-to-implant contact on the mesial and distal aspect of the implant. Marginal bone level expressed in millimeters at the study follow-up visit was compared to values obtained at delivery of permanent restoration i.e. loading (baseline), or within the first 12 months after loading.
Time Frame: Minium of 2 years and a maximum of 8 years of use.
Population: Per protocol population is 142 subjects (259 positions) . For 39 subjects (94 positions) there were no baseline radiographs available for analysis. As a result, a total of 165 positions are included in the analysis of MBL change.
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | ATLANTIS Abutment
Number analyzed (Participants) | 103
Millimeter | -0.30 (0.93)

ADVERSE EVENTS:
Time Frame: Minium of 2 years and a maximum of 8 years
Arm/Group | ATLANTIS Abutment
All-Cause Mortality (participants affected / at risk) | 0/142
Serious Adverse Events (participants affected / at risk) | 0/142
Other Adverse Events (participants affected / at risk) | 0/142

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT02496091/Prot_SAP_000.pdf